CLINICAL TRIAL: NCT04519515
Title: Double Blind Split Face Randomized Placebo Controlled Clinical Trial Investigating Juvederm Vollure for the Correction of Atrophic Facial Scarring
Brief Title: Vollure for the Correction of Atrophic Facial Scarring
Acronym: JVAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Siperstein Dermatology (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JVAS002
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-02

CONDITIONS: Atrophic Scar
Keywords: Hyaluronic Acid Filler; Atrophic Scar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment With Juvederm Vollure Right (Experimental): Injection of Juvederm Vollure on one half of the face, placebo on the other side
  Interventions: Device: Allergan Vollure
- Treatment Juvederm Vollure Left (Experimental): Injection of Juvederm Vollure on one half of the face, placebo on the other side
  Interventions: Device: Allergan Vollure

INTERVENTIONS:
Device: Allergan Vollure — Injection of Allergan Vollure into Atrophic Scars

SUMMARY:
Subjects will be randomized to receive up to 1cc of Juvéderm Vollure on one side of their face and up to 1cc of Saline on the other. On Day 30, this treatment with the same left-right assignment can be repeated. Subjects will return 24-48 hours after their first treatment to fill out questionnaires, take pictures, and to be assessed by blinded evaluators regarding short term adverse events. Subjects will fill out a 30 day subject diary and also return 30 and 90 days after their last treatment to fill out questionnaires, take pictures, complete the Global Aesthetic Improvement Scale (GAIS), and to be assessed on the QGSGS and for long-term adverse events by blinded evaluators. At 12 months, 18 months, and 24 months, the subjects will return to fill out questionnaires, take pictures, and to be assessed by blinded evaluators for long-term efficacy.

DETAILED DESCRIPTION:
Subjects with grades ranging from 4-55 on the Quantitative Global Scarring Grading System (QGSGS)1 will be randomized to receive up to 1cc of Juvéderm Vollure on one side of their face and up to 1cc of Saline on the other. On Day 30, this treatment with the same left-right assignment can be repeated if optimal correction on the active intervention side has not been achieved according to the treating investigator. Subjects will return 24-48 hours after their first treatment to fill out questionnaires, take pictures, and to be assessed by blinded evaluators regarding short term adverse events. Subjects will fill out a 30 day subject diary and also return 30 and 90 days after their last treatment to fill out questionnaires, take pictures, complete the Global Aesthetic Improvement Scale (GAIS), and to be assessed on the QGSGS and for long-term adverse events by blinded evaluators. The subjects will be eligible to receive treatment with Juvéderm Vollure 90 days after their last treatment on the placebo-controlled side if they choose. In addition, at 12 months, 18 months, and 24 months, the subjects will return to fill out questionnaires, take pictures, and to be assessed by blinded evaluators for long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

* In good general health as evidenced by medical history
* For females of reproductive potential: use of highly effective contraception and a negative urine pregnancy test at screening and all injection visits.
* Score of 4-55 on a validated scarring grading system

Exclusion Criteria:

* Subjects with allergies to hyaluronic acid filler, gram positive bacteria or lidocaine.
* Subjects with auto-immune conditions
* Subjects with diabetes
* Subjects with a history of sever anaphylactic reactions
* Subjects with cancer, or other life-threatening medical condition
* Subjects taking anti---coagulants, chemotherapy, immunosuppressive agents, immunomodulatory agents, diuretics, anti---histamines, or anti---inflammatory medications in the 2 weeks prior to the study or who will need to take these medications at any time during the first 120 days of the study.
* Subjects with any scheduled laser, light, or surgical procedures during the study, including dental surgery.
* Subjects who had neuromodulators in the past 6 months or hyaluronic acid fillers in the previous year on the face
* Subjects who at any time had surgery or more permanent fillers in the face such as Bellafill or Radiesse
* Subjects with tattoos or many skin growths on the face that would obscure visualization of the scars
* Subjects with a history of keloid or hypertrophic scar on the face
* Subjects unwilling or unable to sit still while an injector places Juvéderm Vollure in the face
* Subjects unwilling or unable to keep their head still during the photos
* Subjects who are pregnant or nursing
* Female subjects of child-bearing potential unable to take or use some form of birth control
* Subjects with any facial bruising or swelling
* Subjects with current skin infections, tumors, herpes outbreak or dermatitis on the face
* Subjects using skin-irritating topical preparations, pigmenting agents (self-tanning or bleaching creams), in the past two weeks or for the first 120 days of the study on the face
* Any medical condition that in the opinion of the Investigator would make the subject unsuitable for inclusion
* Women who are pregnant or breast feeding, or women of childbearing potential who are not practicing adequate contraception or planning to become pregnant during the study period.
* Study site personnel, close relatives of the study site personnel (e.g. parents, children, siblings, or spouse), employees, or close relatives of employee.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Quantitiative Global Scaring Grading System (QGSGS) score | Baseline to 90 days after last injection
  Difference in the mean QGSGS score from baseline to 90 days after injection in active group. The QGSGS score ranges from 0 to 84 and a higher score signifies a worse condition.

SECONDARY OUTCOMES:
Adverse Events | Baseline to 90 days after last injection
  The difference in number of adverse events from control and active treatment group
Global Aesthetic Improvement Scale (GAIS) | Baseline to 90 days after last injection
  Difference in the mean GAIS score from baseline to 90 days after injection. The scale is a 5 point scale from -1 to 3. A higher score signifies more improvement, a negative score signifies worsening of the condition.
24 Month Global Aesthetic Improvement Scale (GAIS) Results | 24 months after 1st injection
  Difference in the mean GAIS score from baseline to 24 months after injection. The scale is a 5 point scale from -1 to 3. A higher score signifies more improvement, a negative score signifies worsening of the condition.
24 Month Quantitiative Global Scaring Grading System (QGSGS) Results | 24 months after 1st injection
  Difference in the mean QGSGS score from baseline to 24 months after injection. The QGSGS score ranges from 0 to 84 and a higher score signifies a worse condition.
Result of Placebo Group based on the Quantitiative Global Scaring Grading System (QGSGS) | Baseline to 90 days after last injection
  Difference in the mean QGSGS score from baseline to 90 days after injection of placebo group. The QGSGS score ranges from 0 to 84 and a higher score signifies a worse condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Siperstein Dermatology Group, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No